CLINICAL TRIAL: NCT03402646
Title: EFFICACY OF MOBILE PHONE REMINDERS (AND PHOTOVOICE) IN IMPROVING CHILDHOOD IMMUNIZATION UPTAKE AND REDUCING INCIDENCE OF VACCINE-PREVENTABLE DISEASES - A RANDOMIZED CONTROLLED TRIAL AMONG POSTPARTUM MOTHERS AND CAREGIVERS IN NIGERIA
Brief Title: Mobile Phone Reminders (and Photovoice) for Routine Immunization in Nigeria - The MOPING Study
Acronym: MOPING
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: RCSI & UCD Malaysia Campus (Other)
Responsible Party: Principal Investigator, Dr. Surajudeen Abiola Abdulrahman, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: MOPING/V2/07/17
Record Dates: First submitted 2017-12-19; First posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Immunization; Infection
MeSH Terms: conditions — Infections | interventions — Spermine Synthase

STUDY DESIGN:
Intervention Model Description: This will be a single-blind three-arm cluster randomized controlled trial involving post-partum mothers and/or caregivers of infants (age 0-12months) attending immunization clinics in 12 randomly selected Primary Health Care Centres (clusters) across Sokoto, Jigawa, Kano, Ogun, Oyo and Lagos States of Nigeria. Additionally, the investigators will be implementing a photovoice methodology in 6 community clusters (one in each State) involving group discussions between community members (pregnant women in their third trimester, parents/caregivers of infants age 0-12 months), community leaders, service providers and policy makers on benefits of timely immunization and consequences of non-vaccination.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reminder module (SMS and Phone call) (Experimental): Intervention will consist of a "Reminder module" delivered via SMS and telephone calls by an automated, customized software application. This will include standardized SMS reminder 3 days prior to scheduled immunization clinic appointments, telephone call reminders a day prior to scheduled clinic appointment (4 to 6pm) (in addition to standard care - routine paper-based appointment scheduling and counselling by care providers) for routine immunization. Reminders will be provided consistently for all immunization clinic appointments until the child turns 12 months of age.
  Interventions: Behavioral: Reminder module (SMS and Phone call)
- Photovoice (Experimental): In two small groups of 15 participants each per state, purposively selected pregnant women in their third trimester and parents of infants aged 0-12 months in the community, as well as community leaders, service providers and policy makers will be exposed to photographs (taken from other sources) of debilitating consequences of non-immunization, which will form the basis of the group discussions, knowledge sharing and consensus-building sessions, each lasting about 45 minutes to 1 hour. Each community cluster will be linked to a PHC.
  Interventions: Behavioral: Photovoice
- Control (No Intervention): Respondents in control clusters will receive standard care only - comprising routine paper-based appointment scheduling

INTERVENTIONS:
Behavioral: Reminder module (SMS and Phone call) — Same as described under arm/group descriptions
  Arms: Reminder module (SMS and Phone call)
Behavioral: Photovoice — Same as described under arm/group descriptions
  Arms: Photovoice

SUMMARY:
This study aims to implement and test the efficacy of photovoice, Short Messaging Service (SMS) and phone call reminders in improving childhood immunization coverage (uptake, timeliness and completion rates) and reducing incidence of vaccine-preventable diseases (VPDs) among infants in Nigeria

DETAILED DESCRIPTION:
This will be a single-blind three-arm cluster randomized controlled trial involving post-partum mothers and/or caregivers of infants (age 0-12months) attending immunization clinics in 12 randomly selected Primary Health Care Centres (clusters) across Sokoto, Jigawa, Kano, Ogun, Oyo and Lagos States of Nigeria. Additionally, a photovoice methodology will be implemented in 6 community clusters (one in each State) involving group discussions between community members (pregnant women in their third trimester, parents/caregivers of infants age 0-12 months), community leaders, service providers and policy makers on benefits of timely immunization and consequences of non-vaccination. Parent-infant pairs will be followed up for 12 months during which SMS and phone call immunization clinic appointment reminders will be provided to mothers and/or caregivers in intervention arm 1, and photovoice intervention provided at study commencement to participants in intervention arm 2. Respondents in the control group would receive standard care (routine paper-based appointment scheduling alone). The investigators will document and compare immunization uptake (all doses and vaccines), timeliness of receipt and completion rates of scheduled immunization between the three groups, as well as incidence of VPDs between the groups using multivariate statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Mothers/caregivers of healthy infants (age 0 - 12 months) who:

  1. Have a mobile phone access
  2. Received antenatal care and/or delivered their babies in a hospital
  3. Plans to receive immunizations at the selected PHCs
* Purposively-selected community sample of pregnant women in their third trimester, parents/caregivers of infants, providers, community gatekeepers and policy makers

Exclusion Criteria:

1. Parents of infants requiring hospital admission due to significant illness, congenital deformity/malformation and prematurity
2. Foreigners

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1813 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Immunization coverage | 12 months
  Proportion of randomized infants who received birth doses of BCG and OPV (overall), and complete doses of each vaccine as scheduled
Timeliness of receipt of scheduled immunization | 12 months
  Proportion of infants receiving scheduled immunization within 1 week of schedule

SECONDARY OUTCOMES:
Incidence of any childhood vaccine-preventable disease | 12 months
  Risk ratio of vaccine-preventable disease between intervention and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Surajudeen A Abdulrahman, MBBS, PhD, Principal Investigator — RCSI & UCD Malaysia Campus; Niyi Osamiluyi, Study Director — Premier Medical Systems

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276